CLINICAL TRIAL: NCT07393763
Title: Effectiveness of Rectus Sheath Block as an Adjunct to General Anesthesia for Postoperative Pain and Inflammation in Patients Undergoing Midline Incision Laparotomy at RSUP Sanglah
Brief Title: Rectus Sheath Block as an Adjunct to General Anesthesia for Midline Laparotomy Pain
Acronym: RSB-MIDLINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Collaborators: RS Prof. Dr. I.G.N.G Ngoerah (Unknown)
Responsible Party: Principal Investigator, Prema Putra, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022.02.1.0341; 2022.02.1.0341 (Other: Faculty of Medicine, Universitas Udayana); EC-UNUD-82.0-2022 (Other: Research Ethics Committee, Faculty of Medicine, Universitas Udayana)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Abdominal Surgery by Laparotomy
Keywords: Rectus Sheath Block; Midline Laparotomy; Ultrasound-Guided; Opioid Consumption; Numeric Rating Scale; Neutrophil-to-Lymphocyte Ratio; Postoperative Analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Two-arm parallel-group randomized trial comparing general anesthesia alone versus general anesthesia plus bilateral ultrasound-guided rectus sheath block.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were blinded to group assignment. Postoperative pain assessments (NRS) and outcome data collection were performed by an independent assessor who was blinded to allocation. Randomization codes were kept in sealed envelopes and were not disclosed to the assessor until data collection was completed. Data analysis was performed using coded group labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control: General Anesthesia Only (No Intervention): Participants receive standard general anesthesia without rectus sheath block. Postoperative analgesia follows institutional protocol (e.g., PCA morphine and paracetamol).
- Intervention: General Anesthesia + Bilateral Rectus Sheath Block (Experimental): Participants receive standard general anesthesia plus bilateral ultrasound-guided posterior rectus sheath block (single-shot) using bupivacaine 0.25%, 20 mL per side, performed after induction of anesthesia.
  Interventions: Procedure: Ultrasound-guided rectus sheath block

INTERVENTIONS:
Procedure: Ultrasound-guided rectus sheath block — Bilateral posterior rectus sheath block performed under ultrasound guidance after induction of general anesthesia. Single-shot injection of bupivacaine 0.25% (20 mL per side) between the rectus abdominis muscle and posterior rectus sheath.
  Arms: Intervention: General Anesthesia + Bilateral Rectus Sheath Block

SUMMARY:
This study evaluates whether adding an ultrasound-guided rectus sheath block (RSB) to general anesthesia can improve pain control after midline laparotomy. Adult patients undergoing midline incision laparotomy will be randomly assigned to receive either general anesthesia alone or general anesthesia plus bilateral RSB with local anesthetic (bupivacaine 0.25%). After surgery, pain will be assessed using the Numeric Rating Scale (NRS) at 15 minutes, 1 hour, 3 hours, 6 hours, 12 hours, and 24 hours. The study will also compare the time to first opioid request, total opioid use during the first 24 hours after surgery, and changes in inflammation measured by the neutrophil-to-lymphocyte ratio (NLR). The goal is to determine whether RSB can reduce postoperative pain and opioid requirements and help limit postoperative inflammatory response.

DETAILED DESCRIPTION:
This is a double-blind randomized controlled trial conducted in adult patients (18-64 years) undergoing midline incision laparotomy under general anesthesia at Sanglah Hospital. Eligible participants are enrolled consecutively and randomized using permuted block randomization with sealed envelopes into two parallel groups:

Group A (Control): General anesthesia without rectus sheath block.

Group B (Intervention): General anesthesia plus bilateral ultrasound-guided posterior rectus sheath block (RSB) using bupivacaine 0.25%.

Anesthetic management is standardized. Patients receive IV midazolam 0.02 mg/kg as premedication. Induction is performed with propofol 1-2 mg/kg and fentanyl 2 mcg/kg, followed by atracurium 0.5 mg/kg for intubation. Maintenance includes pressure-controlled ventilation (FiO₂ 40%, flow 2 L/min) and propofol infusion 50-150 mcg/kg/min. Intraoperative analgesia is supplemented with fentanyl 0.5 mcg/kg every 45 minutes. Hemodynamics are maintained within 20% of baseline.

RSB technique (Group B): After intubation, the abdominal skin is disinfected. A linear ultrasound probe is placed lateral to the umbilicus to identify the rectus abdominis muscle and posterior rectus sheath. Using an in-plane approach, a 50 mm needle is advanced from lateral to medial until the needle tip lies between the rectus abdominis muscle and posterior rectus sheath. After negative aspiration, 20 mL of bupivacaine 0.25% is injected as a single-shot on one side with aspiration every 3 mL, visualizing separation of the rectus muscle from the posterior sheath. The procedure is then repeated on the contralateral side (bilateral block).

Postoperative management and assessments: Pain is evaluated by an independent observer using the Numeric Rating Scale (NRS 0-10) at T1 (15 minutes in the recovery room), T2 (1 hour), T3 (3 hours), T4 (6 hours), T5 (12 hours), and T6 (24 hours) postoperatively. Postoperative analgesia includes patient-controlled analgesia (PCA) morphine demand-only (1 mg per demand dose) for patients with GCS 15, plus oral paracetamol 500 mg every 6 hours. The time to first opioid request is recorded (minutes), and total morphine consumption during the first 24 hours is collected.

Inflammation assessment: Neutrophil-to-lymphocyte ratio (NLR) is measured from complete blood count (CBC) preoperatively (one day before surgery) and postoperatively (in the recovery room).

Key outcomes include postoperative NRS scores (T1-T6), time to first opioid request, total opioid requirement in the first 24 hours, and perioperative changes in NLR.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-64 years.
* Patients undergoing midline laparotomy incision (incision extending above to below the umbilicus) for digestive, obstetric, or oncology cases (corresponding to T7-T12 dermatomes) under general anesthesia.
* ASA physical status I-III.
* Body mass index (BMI) 18.5-30 kg/m².
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Refusal to participate.
* Infection or wound at the planned block site.
* Decreased level of consciousness.
* Known allergy to local anesthetics or opioids.
* Coagulation disorder.
* History of chronic pain.
* Hyperalgesia.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Intensity (Numeric Rating Scale, NRS) | 15 minutes, 1 hour, 3 hours, 6 hours, 12 hours, and 24 hours after surgery
  Pain intensity measured using the Numeric Rating Scale (0-10; 0 = no pain, 10 = worst imaginable pain) by a blinded assessor.

SECONDARY OUTCOMES:
Time to First Opioid Request | Up to 24 hours after surgery
  Time from arrival in recovery room to first request for opioid analgesia (minutes).
Total Opioid Consumption | 24 hours after surgery
  Total morphine consumption recorded from PCA during the first 24 hours after surgery (mg)
Change in Neutrophil-to-Lymphocyte Ratio (NLR) | Preoperative (1 day before surgery) and postoperative (in recovery room)
  NLR calculated from complete blood count measured preoperatively and postoperatively in the recovery room.
Postoperative Nausea and Vomiting (PONV | Up to 24 hours after surgery
  Incidence of nausea/vomiting within 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: I Made Prema Putra, Principal Investigator — Udayana University
Locations (1):
- Ngoerah Hospital, Denpasar, Bali, Indonesia, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be shared publicly. Data may be considered for sharing upon reasonable request to the principal investigator, subject to institutional and ethics approval